CLINICAL TRIAL: NCT05702723
Title: Building Resiliency Among Caregivers of Curvivors and Metavivors: a Pilot Randomized Trial
Brief Title: Building Resiliency Among Caregivers of Curvivors and Metavivors
Acronym: ForTe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elyse Park, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-357; R21CA273785 (NIH)
Record Dates: First submitted 2023-01-01; First posted 2023-01-27 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Stress; Cancer Diagnosis; Distress, Emotional
Keywords: Stress; Stress Management; Cancer Survivors; Cancer Diagnosis; Emotional Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smart-3RP (Experimental): Survivors-caregivers will be randomized together (dyad), stratified by survivor status: curvivor (participants who have completed curative therapy) or metavivor (participants will metastatic disease), using a random plan generator with 1:1 randomization. Participants will complete study procedures as outlined:
  * Baseline questionnaires.
  * 9 virtual sessions of Smart-3RP.
  * 3-month questionnaires.
  * Optional collections of hair samples at enrollment and 6-month follow-up period to measure cortisol concentration.
  * 6-month questionnaires.
  * Optional exit interview with study staff.
  Interventions: Behavioral: Smart-3RP
- Enhanced Usual Care (Active Comparator): Survivors-caregivers will be randomized together (dyad), stratified by survivor status (curvivor/metavivor), using a random plan generator with 1:1 randomization.
  * Participants will be referred to a 14-week online support group.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Smart-3RP — 9 sessions of mind-body group treatment program via Zoom platform.
  Other Names: Stress Management and Resiliency Training-Relaxation Response Program
  Arms: Smart-3RP
Behavioral: Enhanced Usual Care — 14-week group-based, online support group through CancerCare.org.
  Arms: Enhanced Usual Care

SUMMARY:
The main purpose of this research study is to assess the feasibility and participants' satisfaction of the Stress Management and Resiliency - Relaxation Response Resiliency Program (SMART-3RP) and compare this treatment with SMART-3RP versus referral to a group-based, online support group to see which is better for improving resilience and decreasing distress of participants with cancer and their caregivers.

The name of the study intervention involved in this study is:

Smart-3RP (virtual, mind-body group treatment program).

DETAILED DESCRIPTION:
This pilot, randomized controlled trial assesses the feasibility, acceptability, and efficacy of the Stress Management and Resiliency - Relaxation Response Resiliency Program (SMART-3RP) for improving resiliency and decreasing distress among caregivers and cancer survivors compared to enhanced usual care.

Participants will be randomly assigned into one of the study groups: Smart-3RP versus referral to a group-based, online support group. Randomization means that a participant is placed into a group by chance.

Participation in this study is expected to last about 180 days.

It is expected about 96 people made up of 48 patients and 48 caregivers will take part in this research study.

The National Institutes of Health (NIH) is supporting this research by providing funding.

ELIGIBILITY:
Inclusion Criteria for Patients:

* English speaking adult patients with cancer (18 years or older)
* Treated at MGH, who are either within approximately:

  * 3 months to 3 years after completing potentially curative therapy for cancer diagnosis including surgery, radiation, and/or chemotherapy or other novel therapies (e.g., immunotherapy, biological therapy). Patients can be on long- term maintenance hormonal or biological therapy at the time of enrollment.
  * 6 months to 3 years after diagnosis of metastatic disease with an expected prognosis of >1 year as confirmed by the treating oncology clinician
* Able to identify a caregiver (i.e., spouse/partner or patient-identified family member or friend) who is willing to participate in the study

Exclusion Criteria for Patients:

* Prognosis less than one year as determined by the treating oncology clinician
* Active psychiatric or cognitive comorbidity that prohibits the capacity to provide informed consent as determined by the treating oncology clinician
* Patients without a caregiver who is willing to participate

Inclusion Criteria for Caregivers:

* Adult caregiver (age 18 years or older).
* Identified by the patient as the spouse/partner or family member/friend.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of Enrolled Participants (Feasibility) | At Screening
  Defined as the percent of survivors/caregivers who are eligible enroll, or ≥ 45% enrollment of eligible participants (≥96 enrolled of 213 eligible participants).
Proportion of Intervention Satisfaction (Acceptability) | At 3 months
  Defined as the percent of survivors/caregivers who report overall intervention satisfaction, as 4/5 on Likert scales, or ≥ 75% of participants ( (≥72 of 96 participants).

SECONDARY OUTCOMES:
Proportion of Study Retention (Feasibility) | At 3 months
  Defined as the percent of survivors/caregivers who complete the 3-month follow-up survey, or ≥ 70% of participants (≥67 of 96 participants).
Proportion of Intervention Session Completion (Feasibility) | up to 6 months
  Defined as the percent of survivors/caregivers who attend at least 6 out of 9 intervention sessions, or ≥ 70% of participants (≥67 of 96 participants)
Improvement in Resilience (Exploratory outcome) | At baseline and 3 months
  Assessed by the Current Experiences Scale (CES), a 23-item measure.
Improvement in stress coping (Exploratory outcome) | At baseline and 3 months
  Assessed with the Measure of Current Status (MOCS-A), a 13-item scale.
Health care utilization (exploratory outcome) | At baseline and 6 months
  Having seen a primary care provider in past year
Reduction of Chronic Stress | At baseline and 6 months
  Assessed cortisol level of hair samples

CONTACTS AND LOCATIONS:
Overall Officials: Elyse Park, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Goshe BM, Barata A, Finkelstein-Fox L, Cloutier J, Farnam E, Holmbeck K, Waldron E, Perez GK, Malloy L, Miranda I, Hager W, Horick N, El-Jawahri A, Park E. Study protocol for a pilot randomized trial building resiliency among caregivers of cancer curvivors and metavivors. Contemp Clin Trials Commun. 2025 Jun 19;46:101506. doi: 10.1016/j.conctc.2025.101506. eCollection 2025 Aug. PMID 40606212